CLINICAL TRIAL: NCT00690079
Title: A Phase I, Randomised, Double-blind, Placebo-controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of AZD1386 in Healthy Caucasian Young and Elderly Subjects After Oral Multiple Doses.
Brief Title: Study to Investigate the Safety, Tolerability and Pharmacokinetics of AZD1386
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Rolf Karlsten, MD, PhD Medical Science Director, AstraZeneca R&D Södertälje SE-151 85 Södertälje, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5090C00008; EudraCT No. 2007-005470-31
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2010-12-10 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Pain
Keywords: MAD; Multiple ascending dose; Chronic pain; pain
MeSH Terms: conditions — Chronic Pain; Pain | interventions — AZD1386

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD1386 (Experimental): 7 groups receiving a specified volume of the active component AZD1386 at different points of time.
  Interventions: Drug: AZD1386
- Placebo (Placebo Comparator): 7 groups receiving a specified volume of placebo at different points of time
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD1386 — Oral admin. of doses at 11 days through a 12 days period. Cmax = 16 mikromol/L and AUCmax = 98 mikromol*h/L
  Arms: AZD1386
Drug: Placebo — Oral admin. of doses at 11 days through a 12 days period.
  Arms: Placebo

SUMMARY:
The study is being performed in order to learn more about the safety and tolerability of AZD1386. AZD1386 is primary intended for treatment of chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasians, males or females aged ≥20 and ≤ 45 years or between 65 80 years. Female subjects must be surgically sterile or post-menopausal for at least 12 months prior to the enrolment visit.
* Body Mass Index (BMI) of ≥18 to ≤ 30 kg/m2 and weight of ≥50 to ≤100 kg
* Clinically normal physical findings including heart rate > 45 bpm and laboratory values and normal resting ECG

Exclusion Criteria:

* History of somatic or psychiatric disease/condition, which may interfere with the objectives of the study.
* History of severe allergy/hypersensitivity or symptoms/signs of ongoing allergy/hypersensitivity.
* Subjects with a high decrease in blood pressure within 5 minutes when going from a supine to standing position.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2008-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety AEs and vital signs | During the whole study
ECG-recordings | ECGs (5 minutes) Days 1 and 12. 2 ECGs (5 minutes) Days 3, 6 and 10. 1 ECG (5 minutes) Days 2 and 13.

SECONDARY OUTCOMES:
PK | Days 1, 5 and 12, 12 times each day. Days 4, 6, 8, 10 and 14, once. Days 2, 3, 7, 9, 11 and 13 twice.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Karlsten, Study Director — Emerging Analgesia TA AstraZeneca R&D Södertälje, Sweden; Ray Chetty, Principal Investigator — AstraZeneca Alderly Park1G61 Mereside, Alderly Park, Macclesfeld, Cheshire, England SK104TG
Locations (1):
- Research Site, Macclesfield, Cheshire, United Kingdom